CLINICAL TRIAL: NCT01963364
Title: A Pilot Study Using Magnetic Resonance Imaging to Measure the Effect of Dietary Supplementation With Fructans on Whole Gut Transit Time, Colonic Gas Volume, and Volume Change in Response to a Fructan Challenge
Brief Title: Pilot Study of the Effect of Fructans on Fermentation in the Colon & Transit
Acronym: PERFECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 11072013SCSMRI
Record Dates: First submitted 2013-10-08; First posted 2013-10-16 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2014-01

CONDITIONS: Evidence of Adaptation to Dietary Exposure to Fructans
Keywords: fructans; inulin; oligofructose; colonic fermentation; microbiota; whoe gut transit

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention group (Experimental): All healthy volunteers
  Interventions: Dietary Supplement: Inulin challenge; Dietary Supplement: oligofructose supplement

INTERVENTIONS:
Dietary Supplement: Inulin challenge — On two study days one week apart, fasted participants will consume 500ml of water, flavoured with lime juice, containing 40g inulin.
  Other Names: Orafti HP (Beneo-Orafti, Belgium)
Dietary Supplement: oligofructose supplement — Starting at the end of study day 1, consumption of 5 grams oligofructose coloured with carmine red food dye(<5%), dissolved in a hot drink, twice daily for 6 1/2 days/ 13 doses. The 14th dose of the week is the inulin challenge consumed as part of study day 1.
  Other Names: Orafti P95 (Beneo-Orafti P95, Belgium)

SUMMARY:
Some carbohydrates (complex sugars) which are found in grains, fruit and vegetables, cannot be digested by humans. When eaten they pass through the small bowel to the large bowel, or colon. Some bacteria that live in the colon are able to digest these carbohydrates, and use them as an energy source. This releases energy that humans can absorb, and may have other effects on health as well. The process also releases gases such as hydrogen and methane into the colon, which will eventually be released as flatulence.

There is some evidence in animals, and humans, that changing the carbohydrate content of the diet may increase the numbers of bacteria in the colon that can use this energy source. Recent work has looked at how changes in colon bacteria and carbohydrate in the diet affect transit, the speed at which food and stool moves through the stomach and bowels. This undergraduate project will use techniques in Magnetic Resonance Imaging developed in Nottingham to investigate how a prolonged change in dietary carbohydrate might affect speed of transit through the bowel and gas production in the colon, and whether there is any evidence of a change in the level of signalling chemicals that may affect bowel function.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-55
* Able to give informed consent
* Does not meet criteria for diagnosis of IBS on Rome III questionnaire

Exclusion Criteria:

* Unable to abstain from smoking for the duration of the study (may affect breath hydrogen readings)
* Self-declared vegetarian, vegan or kosher/ halal diet who cannot eat carmine red dye
* Pregnancy declared by candidate
* Female patients during their menstrual period
* History declared by the candidate of pre-existing gastrointestinal disorder, including but not limited to:
* Inflammatory Bowel Disease
* Coeliac Disease
* Pancreatitis
* Gallstone disease (biliary colic, cholecystitis)
* Diverticulitis
* Cancer of the gastrointestinal tract
* Irritable Bowel Syndrome
* Reported history of previous resection of any part of the gastrointestinal tract other than appendix or gallbladder
* Intestinal stoma
* Any medical condition making participation potentially compromising participation in the study e.g. diabetes mellitus, respiratory disease limiting ability to lie in the scanner
* Contraindications for MRI scanning i.e. metallic implants, pacemakers, history of metallic foreign body in eye(s) and penetrating eye injury
* Reported alcohol dependence
* Unable to stop drugs known to alter GI motility including mebeverine, opiates, monoamine oxidase inhibitors, phenothiazines, benzodiazepines, calcium channel antagonists during or in the 2 weeks prior to the test. (Selective serotonin reuptake inhibitors and low dose tricyclic antidepressants will be recorded but will not be an exclusion criteria)
* Antibiotic or probiotic treatment in the past 4 weeks
* Inability to lie flat or exceed scanner limits of weight <120kg
* Poor understanding of English language
* Participation in night shift work the week prior to the study day. Night work is defined as working between midnight and 6.00 AM
* Strenuous exercise greater than 10 hours per week (i.e. no competition training the week prior to the study).
* Participation in any medical trials for the past 3 months
* Anyone who in the opinion of the investigator is unlikely to be able to comply with the protocol e.g. cognitive dysfunction, chaotic lifestyle related to substance abuse

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2013-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in whole gut transit time after one week (measured in hours) calculated using MRI marker capsule technique | Difference (Delta) between baseline and after one week of intervention
  5 markers pills will be swallowed 24 hours before MRI scanning. Each pill will be given a score 0-9 based on the colonic segment where it is located. The weighted mean of these scores will be the geometric centre. Previous validation allows a transit time to be calculated from the geometric centre.

SECONDARY OUTCOMES:
Change in fasting colonic volume | Baseline and after one week of intervention
  Calculated from segmentation on MRI scans
Change in colonic volume 8 hours after ingestion of 40 grams inulin dissolved in 500ml water flavoured with lime juice, measured in millilitres | Baseline and after one week of intervention
  Calculated from segmentation on MRI scans
Change in fasting colonic gas volume, measured in millilitres | Baseline and after one week of intervention
  Measured using MRI segmentation technique
Change in colonic gas volume 8 hours after ingestion of 40 grams inulin dissolved in 500ml water flavoured with lime juice, measured in millilitres | Baseline and after one week of intervention
  Calculated from segmentation on MRI scans
Change in breath hydrogen concentration, measured in parts per million before, 4 hours after, and 8 hours after ingestion of 40 grams inulin | Baseline and after one week of intervention
Change in faecal 5-HIAA concentration in μmol/g | baseline and after one week of intervention
  measured by high performance liquid chromatography

OTHER OUTCOMES:
Presence of clinically important digestive symptoms during study day or intervention week | one week of intervention
  * We will measure 4 symptoms from a previously validated questionnaire on a scale of 0 (none), 1 (mild/ distinct but negligible), 2 (moderate/ annoying), 3 (severe/ disabling), and also on a Visual Analogue Scale (0-100)
  * Symptoms include abdominal pain, bloating, gas/flatulence, and diarrhoea.
  * We will define clinically important symptoms as a composite score of 3 or more at any time point or on any day.

CONTACTS AND LOCATIONS:
Overall Officials: Robin C Spiller, MD, Principal Investigator — University of Nottingham; Giles Major, MD, Principal Investigator — University of Nottingham; Luca Marciani, PhD, Principal Investigator — University of Nottingham
Locations (2):
- United Kingdom (2):
  - Sir Peter Mansfield Magnetic Resonance Centre, Nottingham
  - Nottingham Digestive Diseases Centre, Nottingham

REFERENCES:
- See also: The unit website — http://www.nddcbru.org.uk